CLINICAL TRIAL: NCT02208037
Title: A Multi-center Phase II Trial Randomizing Novel Approaches for Graft-versus-Host Disease Prevention Compared to Contemporary Controls (BMT CTN #1203; Progress I)
Brief Title: Novel Approaches for Graft-versus-Host Disease Prevention Compared to Contemporary Controls (BMT CTN 1203)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BMTCTN1203; U01HL069294 (NIH)
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2017-12

CONDITIONS: Acute Leukemia; Chronic Myelogenous Leukemia; Myelodysplasia; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Hodgkin's Lymphoma
Keywords: Acute Lymphoblastic Leukemia/Lymphoma; Acute Myelogenous Leukemia; Mantel-Cell Lymphoma; Hematopoietic Transplant; GVHD Prophylaxis
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Refractory, with Excess of Blasts; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Tacrolimus; Methotrexate; Cyclophosphamide; Maraviroc; Bortezomib; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tacrolimus/Methotrexate/Bortezomib (Experimental): Participants will receive specified dosage of three different GVHD prophylaxis agents: Tacrolimus, Methotrexate, and Bortezomib.
  Interventions: Drug: Tacrolimus (ARM with Methotrexate); Drug: Methotrexate (ARM with Bortezomib); Drug: Bortezomib
- Tacrolimus/Methotrexate/Maraviroc (Experimental): Participants will receive specified dosage of three different GVHD prophylaxis agents: Tacrolimus, Methotrexate, and Maraviroc.
  Interventions: Drug: Tacrolimus (ARM with Methotrexate); Drug: Methotrexate (ARM with Maraviroc); Drug: Maraviroc
- Tacrolimus/MMF/Cyclophosphamide (Experimental): Participants will receive specified dosage of three different GVHD prophylaxis agents: Tacrolimus, Mycophenolate Mofetil (MMF), and Cyclophosphamide.
  Interventions: Drug: Tacrolimus (ARM with MMF and Cyclophosphamide); Drug: Mycophenolate mofetil; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Tacrolimus (ARM with Methotrexate) — Tacrolimus will be given orally at a dose of 0.05 mg/kg or intravenously at a dose of 0.03 mg/kg starting Day -3. The dose of tacrolimus may be rounded to the nearest 0.5 mg for oral formulations. Subsequent dosing will be based on blood levels. The dose should be adjusted accordingly to maintain a suggested level of 5-15 ng/mL. If patients are on medications which alter the metabolism of tacrolimus (e.g. azoles), the initial starting dose and subsequent doses should be altered as per institutional practices. Tacrolimus taper can be initiated at a minimum of 90 days post HSCT if there is no evidence of active GVHD. The rate of tapering will be done according institutional practices but patients should be off tacrolimus by Day 180 post HSCT if there is no evidence of active GVHD.
  Other Names: Prograf®; FK506
  Arms: Tacrolimus/Methotrexate/Bortezomib; Tacrolimus/Methotrexate/Maraviroc
Drug: Tacrolimus (ARM with MMF and Cyclophosphamide) — Tacrolimus will be given orally at a dose of 0.05 mg/kg or intravenously at a dose of 0.03 mg/kg starting Day +5. Serum levels of tacrolimus will be measured at Day 7 and then should be checked weekly thereafter, and the dose adjusted accordingly to maintain a suggested level of 5-15 ng/mL. Tacrolimus taper can be initiated at a minimum of 90 days post HSCT if there is no evidence of active GVHD. The rate of tapering will be done according to institutional practices but patients should be off tacrolimus by Day 180 post HSCT if there is no evidence of active GVHD.
  Other Names: Prograf®; FK506
  Arms: Tacrolimus/MMF/Cyclophosphamide
Drug: Methotrexate (ARM with Maraviroc) — Methotrexate will be administered, per institutional practices, at the doses of 15 mg/m2 IV bolus on Day +1, and 10 mg/m2 IV bolus on Days +3, +6 and +11 after hematopoietic stem cell infusion. The Day +1 dose of methotrexate will be given at least 24 hours after the hematopoietic stem cell infusion and at least 30 minutes after the first dose of maraviroc. Dose reduction of MTX due to worsening creatinine clearance after initiation of conditioning regimen, high serum levels or development of oral mucositis is allowed according to institutional practices.
  Other Names: MTX
  Arms: Tacrolimus/Methotrexate/Maraviroc
Drug: Methotrexate (ARM with Bortezomib) — Methotrexate will be administered, per institutional practices, at the doses of 15 mg/m2 IV bolus on Day +1, and 10 mg/m2 IV bolus on Days +3, +6 and +11 after hematopoietic stem cell infusion. The Day +1 dose of methotrexate will be given at least 24 hours after the hematopoietic stem cell infusion and at least 30 minutes after the first dose of bortezomib. Dose reduction of MTX due to worsening creatinine clearance after initiation of conditioning regimen, high serum levels or development of oral mucositis is allowed according to institutional practices.
  Other Names: MTX
  Arms: Tacrolimus/Methotrexate/Bortezomib
Drug: Maraviroc — Maraviroc will be dosed at 300 mg orally twice a day and will start on Day -3 prior to hematopoietic stem cell infusion, and continue until Day 30 post HSCT. If the patient requires a two-day stem cell infusion, maraviroc treatment will end 30 days after the first infusion day.
  Other Names: Selzentry®
  Arms: Tacrolimus/Methotrexate/Maraviroc
Drug: Bortezomib — Bortezomib will be administered at the dose of 1.3 mg/m2 based upon actual body weight (ABW) as an approximately 3-5 second IV push on Days +1, +4, and +7 after hematopoietic stem cell infusion. There must be at least 72 hours between each dose of bortezomib. Subcutaneous administration of bortezomib is not allowed on this protocol.
  Other Names: Velcade®
  Arms: Tacrolimus/Methotrexate/Bortezomib
Drug: Mycophenolate mofetil — MMF will be given at a dose of 15 mg/kg three times a day (TID) based upon ABW with the maximum total daily dose not to exceed 3 grams (1g TID, IV or PO). MMF prophylaxis will start Day 5 and discontinue after the last dose on Day 35, or may be continued if active GVHD is present.
  Other Names: Cellcept®
  Arms: Tacrolimus/MMF/Cyclophosphamide
Drug: Cyclophosphamide — Hydration prior to cyclophosphamide may be given according to institutional standards.
  Mesna will be given in divided doses IV 30 min pre- and at 3, 6, and 8 hours post-cyclophosphamide or administered per institutional standards. Mesna dose will be based on the cyclophosphamide dose being given. The total daily dose of Mesna is equal to 80% of the total daily dose of cyclophosphamide.
  Cyclophosphamide [50 mg/kg ideal body weight (IBW); if ABW < IBW, use ABW] will be given on Day 3 post-transplant (between 60 and 72 hours after the start of the HSCT) and on Day 4 post-transplant (approximately 24 hours after Day 3 cyclophosphamide). Cyclophosphamide will be given as an IV infusion over 1-2 hours (depending on volume).
  Other Names: Cytoxan®
  Arms: Tacrolimus/MMF/Cyclophosphamide

SUMMARY:
Acute Graft-versus-Host-Disease (GVHD) is an important cause of morbidity and mortality after allogeneic hematopoietic stem cell transplantation (HSCT). This study aims to determine if any of three new GVHD prophylaxis approaches improves the rate of GVHD and relapse free survival at one year after transplant compared to the current standard prophylaxis regimen.

DETAILED DESCRIPTION:
GVHD is a complication that can occur after a bone marrow or stem cell transplant. The transplant recipient's body is attacked by the newly introduced cells. Only about 40% of patients with acute GVHD have durable responses when treated with corticosteroid therapy. A strategy that helps fewer people suffer from GVHD, without other adverse effects, would be an effective approach to improve survival after allogeneic transplantation.

GVHD incidence can be decreased with various treatment plans. Early transplants were done using post-transplant methotrexate to prevent GVHD. Another drug, cyclosporine, was later shown to work better than methotrexate. Then doctors discovered that the combined use of cyclosporine and methotrexate worked even better than either agent alone. More recently, other calcineurin-inhibitors, such as tacrolimus have been developed as GVHD prophylactic agents due to favorable toxicity profiles in comparison with cyclosporine. Studies have been conducted to compare available treatment combinations for related and unrelated donors. The combination of tacrolimus/methotrexate remains a standard for GVHD prophylaxis.

However, improved GVHD prophylaxis remains a significant clinical need in HSCT. The current clinical trial will test three novel GVHD prophylaxis approaches: tacrolimus/methotrexate and bortezomib (Tac/MTX/Bort), tacrolimus/methotrexate and maraviroc (Tac/MTX/MVC) and tacrolimus/mycophenolate mofetil and cyclophosphamide (Tac/MMF/Cy). This randomized Phase II clinical trial will compare each intervention arm with a Tac/MTX control.

This study will enroll people who have a cancer of the blood or lymph glands and a stem cell transplant is a treatment option. The study will take at least two years and will include 270 participants - 90 participants in each of three treatment groups. The purpose of this study is to compare three combinations of medications to see whether one or more of them are better than the current standard of care (Tacrolimus/Methotrexate) to prevent GVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years (patient is older than 18.0 and less than 76.0 years old)
2. Patients with acute leukemia, chronic myelogenous leukemia or myelodysplasia with no circulating blasts and with less than 5% blasts in the bone marrow.
3. Patients with chronic lymphocytic leukemia/small lymphocytic lymphoma, follicular, marginal zone, diffuse large B-cell, Hodgkin's Lymphoma,or mantle cell lymphoma with chemosensitive disease at time of transplantation
4. Planned reduced intensity conditioning regimen (see eligible regimens in Table 2.4a)
5. Patients must have a related or unrelated peripheral blood stem cell donor as follows:

   1. Sibling donor must be a 6/6 match for HLA-A and -B at intermediate (or higher) resolution, and -DRB1 at high resolution using DNA-based typing, and must be willing to donate peripheral blood stem cells and meet institutional criteria for donation.
   2. Unrelated donor must be a 7/8 or 8/8 match at HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing. Unrelated donor must be willing to donate peripheral blood stem cells and be medically cleared to donate stem cells according to National Marrow Donor Program (NMDP) criteria.
6. Cardiac function: Ejection fraction at rest ≥ 45%
7. Estimated creatinine clearance greater than 50 mL/minute (using the Cockcroft-Gault formula and actual body weight)
8. Pulmonary function: Diffusing capacity of the lung for carbon monoxide (DLCO) ≥ 40% (adjusted for hemoglobin) and forced expiratory volume in one second (FEV1) ≥ 50%
9. Liver function: total bilirubin < 1.5 x the upper limit of normal and alanine aminotransferase (ALT)/aspartate aminotransferase (AST) < 2.5x the upper normal limit. Patients who have been diagnosed with Gilbert's Disease are allowed to exceed the defined bilirubin value of 1.5x the upper limit of normal.
10. Female subjects (unless postmenopausal for at least 1 year before the screening visit, or surgically sterilized), agree to practice two (2) effective methods of contraception at the same time, or agree to completely abstain from heterosexual intercourse, from the time of signing the informed consent through 12 months post transplant (see Section 2.6.4 for definition of postmenopausal).
11. Male subjects (even if surgically sterilized), of partners of women of childbearing potential must agree to one of the following: practice effective barrier contraception (see Section 2.6.4 for list of barrier methods), or abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post transplant.
12. Signed informed consent

Exclusion Criteria:

1. Prior allogeneic transplant
2. Karnofsky Performance Score < 70%
3. Active central nervous system (CNS) involvement by malignant cells
4. Patients with uncontrolled bacterial, viral or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment.
5. Presence of fluid collection (ascites, pleural or pericardial effusion) that interferes with methotrexate clearance or makes methotrexate use contraindicated
6. Patients with transformed lymphoma (e.g., Richters transformation arising in follicular lymphoma or chronic lymphocytic leukemia)
7. Patients seropositive for the human immunodeficiency virus (HIV)
8. Patient with active Hepatitis B or C determined by serology and/or nucleic acid amplification tests (NAAT)
9. Patients with hypersensitivity to bortezomib, boron or mannitol
10. Patients with ≥ grade 2 sensory peripheral neuropathy
11. Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure (see Appendix D), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
12. Female patients who are lactating or pregnant
13. Patients with a serious medical or psychiatric illness likely to interfere with participation in this clinical study
14. Patients with prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously will not be allowed unless approved by the Protocol Officer or one of the Protocol Chairs.
15. Planned use of anti-thymocyte globulin (ATG) or alemtuzumab in conditioning regimen.
16. Planned post-transplant therapy, including use of tyrosine-kinase inhibitors (TKI).
17. Inability to withhold agents that may interact with hepatic cytochrome P450 enzymes (CYP3A4), or glutathione S-transferases involved in bortezomib and/or busulfan metabolism during day -5 through day +7. It is acceptable to use alternative non-interacting medications during this period, and then resume prior medications.
18. Patients with secondary acute myeloid leukemia arising from myeloproliferative disease, including Chronic myelomonocytic leukemia (CMML), with evidence of active myeloproliferative features or myelofibrosis in the background.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2014-08; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (30):
- United States (30):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - BMT Program at Northside Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Westwood, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute/Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute/Brigham & Women's, Boston, Massachusetts
  - Karmanos Cancer Institute/BMT, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, Manhattan, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas/MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - University of Utah Med School, Salt Lake City, Utah
  - Virginia Commonwealth University MCV Hospitals, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Derived] Bolanos-Meade J, Reshef R, Fraser R, Fei M, Abhyankar S, Al-Kadhimi Z, Alousi AM, Antin JH, Arai S, Bickett K, Chen YB, Damon LE, Efebera YA, Geller NL, Giralt SA, Hari P, Holtan SG, Horowitz MM, Jacobsohn DA, Jones RJ, Liesveld JL, Logan BR, MacMillan ML, Mielcarek M, Noel P, Pidala J, Porter DL, Pusic I, Sobecks R, Solomon SR, Weisdorf DJ, Wu J, Pasquini MC, Koreth J. Three prophylaxis regimens (tacrolimus, mycophenolate mofetil, and cyclophosphamide; tacrolimus, methotrexate, and bortezomib; or tacrolimus, methotrexate, and maraviroc) versus tacrolimus and methotrexate for prevention of graft-versus-host disease with haemopoietic cell transplantation with reduced-intensity conditioning: a randomised phase 2 trial with a non-randomised contemporaneous control group (BMT CTN 1203). Lancet Haematol. 2019 Mar;6(3):e132-e143. doi: 10.1016/S2352-3026(18)30221-7. PMID 30824040

RESULTS

PARTICIPANT FLOW:
Groups:
- Tacrolimus/Methotrexate/Bortezomib: Participants will receive a GVHD prophylactic regimen of three agents: Tacrolimus, Methotrexate, and Bortezomib.
- Tacrolimus/Methotrexate/Maraviroc: Participants will receive a GVHD prophylactic regimen of three agents: Tacrolimus, Methotrexate, and Maraviroc.
- Tacrolimus/MMF/Cyclophosphamide: Participants will receive a GVHD prophylactic regimen of three agents: Tacrolimus, Mycophenolate Mofetil (MMF), and Cyclophosphamide.
Period: Overall Study
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Started | 93 | 93 | 93
Completed | 89 | 92 | 92
Not Completed | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide | Total
Number analyzed (Participants) | 89 | 92 | 92 | 273
Age, Continuous [Median (Full Range); unit: years] | 64 [28 to 76] | 64 [24 to 74] | 64 [25 to 75] | 64 [24 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 37 | 30 | 98
  Male | 58 | 55 | 62 | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 7 | 11
  Not Hispanic or Latino | 85 | 86 | 81 | 252
  Unknown or Not Reported | 3 | 3 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 3 | 7
  White | 79 | 81 | 82 | 242
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 4 | 7 | 5 | 16
HCT-CI Comorbidity Index [Count of Participants; unit: Participants] — The HCT-CI is a measure of comorbidities present in hematopoietic cell transplant patients. It is scored on an integer-valued scale from 0-29, with greater values indicating greater levels of comorbidity.
  Participants
    0 | 24 | 18 | 26 | 68
    1-2 | 31 | 37 | 27 | 95
    3 or greater | 34 | 37 | 39 | 110
Karnofsky Performance Score [Count of Participants; unit: Participants] — KPS describes patient-perceived global quality of life and functioning on a scale of 0-100.
  100: No evidence of disease; 90: Normal activity. Minor signs or symptoms of disease; 80: Normal activity with effort. Some signs or symptoms of disease; 70: Cares for self. Unable to continue normal activity; 60: Needs occasional assistance, but cares for most personal needs; 50: Needs considerable assistance and medical care; 40: Disabled. Needs special care and assistance; 30: Severely disabled. Hospital admission indicated; 20: Very sick. Active supportive therapy needed; 10: Moribund; 0: Dead
  Participants
    100 | 13 | 10 | 11 | 34
    90 | 39 | 39 | 42 | 120
    80 | 29 | 27 | 28 | 84
    70 | 8 | 16 | 11 | 35
HLA Matching and Donor Type [Count of Participants; unit: Participants] — For related donors, HLA matching was performed on 6 markers using HLA-A and -B at intermediate resolution and -DRB1 at high resolution. For unrelated donors, matching was performed on 8 markers using HLA-A, -B, -C and -DRB1 at high resolution.
  Participants
    Matched Sibling (6/6) | 29 | 33 | 29 | 91
    Matched Other Relative (6/6) | 1 | 1 | 4 | 6
    Matched Unrelated (8/8) | 53 | 48 | 50 | 151
    Mismatched Unrelated (7/8) | 6 | 10 | 9 | 25
Primary Diagnosis [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia (AML) | 46 | 49 | 49 | 144
  Acute Lymphoblastic Leukemia (ALL) | 12 | 11 | 8 | 31
  Chronic Myelogeneous Leukemia (CML) | 2 | 2 | 3 | 7
  Chronic Lymphocytic Leukemia (CLL) | 2 | 3 | 0 | 5
  Myelodysplastic Syndrome (MDS) | 16 | 15 | 17 | 48
  Follicular Lymphoma | 3 | 6 | 5 | 14
  Diffuse Large B-Cell Lymphoma | 4 | 1 | 7 | 12
  Mantle Cell Lymphoma | 4 | 4 | 1 | 9
  Hodgkin's Lymphoma | 0 | 1 | 2 | 3
Time from Diagnosis to Transplant [Median (Full Range); unit: months] | 7.1 [2.1 to 110.3] | 6.3 [2.0 to 122.5] | 7.4 [2.1 to 139.4] | 7.1 [2.0 to 139.4]
Donor/Recipient Sex Matching [Count of Participants; unit: Participants]
  Male donor / Male Recipient | 44 | 39 | 43 | 126
  Male donor / Female Recipient | 19 | 18 | 20 | 57
  Female donor / Male Recipient | 14 | 16 | 19 | 49
  Female donor / Female Recipient | 12 | 19 | 10 | 41
Donor/Recipient Cytomegalovirus (CMV) Status [Count of Participants; unit: Participants]
  Donor Positive / Recipient Positive | 29 | 28 | 25 | 82
  Donor Positive / Recipient Negative | 4 | 19 | 7 | 30
  Donor Negative / Recipient Positive | 25 | 19 | 26 | 70
  Donor Negative / Recipient Negative | 31 | 26 | 34 | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With GVHD/Relapse or Progression-free Survival (GRFS)
Description: GRFS is defined as being free of grade III-IV acute GVHD onset, chronic GVHD onset requiring systemic immunosuppressive therapy, disease relapse or progression, and death from any cause.
Time Frame: 1 Year Post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
percentage of participants | 35.5 [27.2 to 43.9] | 27.2 [19.9 to 35.0] | 44.1 [35.3 to 52.4]

2. Secondary Outcome: Percentage of Participants With Grade II-IV Acute GVHD
Description: Acute GVHD is graded according to the scoring system proposed by Przepiorka et al.1995:
  Skin stage:
  0: No rash
  1. Rash <25% of body surface area
  2. Rash on 25-50% of body surface area
  3. Rash on > 50% of body surface area
  4. Generalized erythroderma with bullous formation
  Liver stage (based on bilirubin level)*:
  0: <2 mg/dL
  1. 2-3 mg/dL
  2. 3.01-6 mg/dL
  3. 6.01-15.0 mg/dL
  4. >15 mg/dL
  GI stage*:
  0: No diarrhea or diarrhea <500 mL/day
  1. Diarrhea 500-999 mL/day or persistent nausea with histologic evidence of GVHD
  2. Diarrhea 1000-1499 mL/day
  3. Diarrhea >1500 mL/day
  4. Severe abdominal pain with or without ileus * If multiple etiologies are listed for liver or GI, the organ system is downstaged by 1.
  GVHD grade:
  0: All organ stages 0 or GVHD not listed as an etiology I: Skin stage 1-2 and liver and GI stage 0 II: Skin stage 3 or liver or GI stage 1 III: Liver stage 2-3 or GI stage 2-4 IV: Skin or liver stage 4
Time Frame: Day 180 Post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
percentage of participants | 26 [19 to 34] | 32 [24 to 40] | 27 [20 to 35]

3. Secondary Outcome: Percentage of Participants With Grade III-IV Acute GVHD
Description: Acute GVHD is graded according to the scoring system proposed by Przepiorka et al.1995:
  Skin stage:
  0: No rash
  1. Rash <25% of body surface area
  2. Rash on 25-50% of body surface area
  3. Rash on > 50% of body surface area
  4. Generalized erythroderma with bullous formation
  Liver stage (based on bilirubin level)*:
  0: <2 mg/dL 1.2-3 mg/dL 2.3.01-6 mg/dL 3.6.01-15.0 mg/dL 4.>15 mg/dL
  GI stage*:
  0: No diarrhea or diarrhea <500 mL/day
  1. Diarrhea 500-999 mL/day or persistent nausea with histologic evidence of GVHD
  2. Diarrhea 1000-1499 mL/day
  3. Diarrhea >1500 mL/day
  4. Severe abdominal pain with or without ileus * If multiple etiologies are listed for liver or GI, the organ system is downstaged by 1.
  GVHD grade:
  0: All organ stages 0 or GVHD not listed as an etiology I: Skin stage 1-2 and liver and GI stage 0 II: Skin stage 3 or liver or GI stage 1 III: Liver stage 2-3 or GI stage 2-4 IV: Skin or liver stage 4
Time Frame: Day 180 Post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
percentage of participants | 8 [4 to 13] | 9 [4 to 14] | 2 [0 to 5]

4. Secondary Outcome: Percentage of Participants With Chronic GVHD
Description: Chronic GVHD is classified per 2005 NIH Consensus Criteria (Filipovich et al. 2005) into categories of severity: none, mild, moderate, and severe. Occurrence of chronic GVHD is defined as the occurrence of mild, moderate, or severe chronic GVHD per this classification.
Time Frame: 1 Year Post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
percentage of participants | 39 [30 to 48] | 43 [35 to 52] | 28 [20 to 36]

5. Secondary Outcome: Percentage of Participants With Chronic GVHD Requiring Immunosupressive Therapy
Description: Chronic GVHD is classified per 2005 NIH Consensus Criteria (Filipovich et al. 2005) into categories of severity: none, mild, moderate, and severe. Occurrence of chronic GVHD is defined as the occurrence of mild, moderate, or severe chronic GVHD per this classification. This endpoint considers the occurrence of chronic GVHD that necessitated initiation of immunosuppressive therapy for treatment.
Time Frame: 1 Year Post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
percentage of participants | 29 [22 to 38] | 33 [25 to 41] | 22 [15 to 30]

6. Secondary Outcome: Percentage of Participants With Disease Relapse or Progression
Description: Relapse is defined by either morphological or cytogenetic evidence of acute leukemia or MDS consistent with pretransplant features, or radiologic evidence of lymphoma. Progression of disease applies to patients with lymphoproliferative diseases (lymphoma or chronic lymphocytic leukemia) not in remission prior to transplantation and is defined as increase in size of prior sites of disease or evidence of new sites of disease.
Time Frame: 1 Year Post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
percentage of participants | 24 [17 to 32] | 31 [23 to 39] | 28 [21 to 37]

7. Secondary Outcome: Percentage of Participants With Transplant-Related Mortality (TRM)
Description: TRM is defined as death without prior disease relapse or progression.
Time Frame: 1 Year Post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
percentage of participants | 17 [11 to 24] | 16 [10 to 23] | 11 [6 to 17]

8. Secondary Outcome: Percentage of Participants With Disease-free Survival
Description: Disease-free survival is defined as being alive and free of disease relapse or progression.
Time Frame: 1 Year Post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
percentage of participants | 58 [49 to 66] | 56 [47 to 64] | 60 [51 to 68]

9. Secondary Outcome: Percentage of Participants With GVHD-free Survival
Description: GVHD-free survival is defined as being alive without previous onset of Grade III-IV acute GVHD or chronic GVHD requiring immunosuppressive therapy.
Time Frame: 1 Year Post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
percentage of participants | 43 [34 to 52] | 34 [26 to 42] | 53 [44 to 61]

10. Secondary Outcome: Percentage of Participants With Overall Survival
Time Frame: 1 Year Post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
percentage of participants | 68 [59 to 76] | 66 [57 to 74] | 71 [63 to 78]

11. Secondary Outcome: Percentage of Participants With Neutrophil Recovery
Description: Neutrophil recovery is defined as achieving an absolute neutrophil count (ANC) ≥ 500/mm^3 for three consecutive measurements on three different days.
Time Frame: Days 28 and 100 Post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
percentage of participants
  Day 28 | 94 [89 to 98] | 93 [89 to 97] | 95 [90 to 98]
  Day 100 | 96 [91 to 99] | 95 [90 to 98] | 98 [94 to 100]

12. Secondary Outcome: Percentage of Participants With Platelet Recovery
Description: Platelet recovery is defined as the first day of a sustained platelet count >20,000/mm^3 with no platelet transfusion in the preceding seven days.
Time Frame: Days 60 and 100 Post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
percentage of participants
  Day 60 | 91 [85 to 96] | 92 [87 to 96] | 90 [84 to 95]
  Day 100 | 91 [85 to 96] | 92 [87 to 96] | 96 [91 to 99]

13. Secondary Outcome: Donor Cell Engraftment
Description: Donor cell engraftment will be assessed with donor/recipient chimerism. Chimerism may be evaluated in bone marrow, whole blood, or CD3 fractions. Full donor chimerism is defined as the presence of ≥ 95% of donor cells as a proportion of total cells. Mixed chimerism is defined as the presence of donor cells, as a proportion of total cells, of < 95% but > 5% in the bone marrow or peripheral blood. Full and mixed chimerism will be evidence of donor cell engraftment. Donor cells of ≤ 5% will be considered as graft rejection.
Time Frame: Days 28 and 100 Post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
Participants
  Day 28: Full Chimerism | 58 | 56 | 64
  Day 28: Mixed Chimerism | 11 | 10 | 8
  Day 28: Graft Rejection | 1 | 1 | 2
  Day 28: Dead | 2 | 4 | 0
  Day 28: No Assay Performed | 17 | 21 | 18
  Day 100: Full Chimerism | 63 | 56 | 62
  Day 100: Mixed Chimerism | 14 | 17 | 13
  Day 100: Graft Rejection | 5 | 3 | 3
  Day 100: Dead | 4 | 10 | 5
  Day 100: No Assay Performed | 3 | 6 | 9

14. Secondary Outcome: Primary Cause of Death
Time Frame: 1 Year Post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
Number analyzed (Participants) | 89 | 92 | 92
Participants
  Recurrence/Persistence | 11 | 12 | 15
  Acute GVHD | 3 | 7 | 2
  Chronic GVHD | 2 | 1 | 1
  Infection | 4 | 7 | 4
  Organ Failure | 2 | 2 | 2
  Hemorrhage | 1 | 0 | 1
  Interstitial Pneumonia | 1 | 0 | 1
  Adult Respiratory Distress Syndrome | 2 | 1 | 0
  Metastatis Breast Cancer | 1 | 0 | 0
  Squamous Cell Carcinoma | 1 | 0 | 0
  Toxicity - Not Specified | 0 | 1 | 0
  Still Alive | 61 | 61 | 66

ADVERSE EVENTS:
Time Frame: Up to 1 Year Post-transplant
Arm/Group | Tacrolimus/Methotrexate/Bortezomib | Tacrolimus/Methotrexate/Maraviroc | Tacrolimus/MMF/Cyclophosphamide
All-Cause Mortality (participants affected / at risk) | 30/93 | 31/93 | 27/93
Serious Adverse Events (participants affected / at risk) | 21/93 | 14/93 | 12/93
Other Adverse Events (participants affected / at risk) | 0/93 | 0/93 | 0/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus/Methotrexate/Bortezomib (N=93) | Tacrolimus/Methotrexate/Maraviroc (N=93) | Tacrolimus/MMF/Cyclophosphamide (N=93)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Anorectal cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02208037/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT02208037/SAP_001.pdf